CLINICAL TRIAL: NCT01937442
Title: A Phase 1, Open-label Study to Evaluate the Pharmacokinetics of Thalidomide Following Multiple Oral Dosing in Subjects With Multiple Myeloma
Brief Title: Pharmacokinetic Study of Thalidomide in Subjects With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CC-2001-CP-001; 2012-005529-62 (EudraCT Number)
Record Dates: First submitted 2013-09-04; First posted 2013-09-09 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Pharmacokinetics; Thalidomide
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thalidomide Celgene™ 200mg once daily (Experimental): 5-day period of thalidomide treatment
  Interventions: Drug: Thalidomide Celgene™

INTERVENTIONS:
Drug: Thalidomide Celgene™ — 200mg once daily and by mouth

SUMMARY:
Objective of this study is to characterize the steady-state pharmacokinetics (PK) of thalidomide when given orally as monotherapy to subjects with multiple myeloma.

DETAILED DESCRIPTION:
This is an open-label, PK study in multiple myeloma subjects who are currently receiving thalidomide-containing therapy or are newly diagnosed. The study will consist of a screening phase, a baseline phase, a PK phase with a 5-day period of thalidomide treatment (200 mg/day), and an end-of-study evaluation on Day 6. Subjects will have frequent blood samples drawn for PK assessments on Days 5 and 6 in an inpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ at 18 the time of signing the informed consent document.
* Documented diagnosis of multiple myeloma and receiving thalidomide containing therapy or initiating thalidomide-containing therapy.
* Subjects must agree to temporally discontinue all antimyeloma therapies other than the study drug (thalidomide) at least 7 days prior to the PK phase (Day 1) and through post study procedures on Day 6.
* All Females of Child Bearing Potential (FCBP) and male subjects must be counseled about pregnancy precautions and risks of fetal exposure.
* Females of childbearing potential (FCBP) must:

  1. Have two negative pregnancy tests as verified by the study doctor prior to starting study therapy. She must agree to ongoing pregnancy testing during the course of the study, and after end of study therapy. This applies even if the subject practices true abstinence from heterosexual contact.
  2. Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis) or agree to use, and be able to comply with, effective contraception without interruption, 28 days prior to starting study drug, during the study therapy (including dose interruptions), and for 28 days after discontinuation of study therapy.
* All other females must had either a hysterectomy or bilateral oophorectomy at least 6 months before screening (proper documentation required) OR been naturally postmenopausal for at least 24 consecutive months (i.e. who has not had menses at any time in the preceding 24 consecutive months). For this study, in subjects who are postmenopausal, estradiol level must be <30 pg/mL and plasma FSH must be >40 IU/L at screening.
* Males (including those who have had a vasectomy):

  1. Must practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 28 days following study drug discontinuation, even if he has undergone a successful vasectomy.
  2. Must agree to not donate semen and sperm during study drug therapy and for 4 weeks after end of study drug therapy.
* All subjects must also be counseled against sharing thalidomide and donating blood during and within 4 weeks of discontinuing thalidomide therapy

Exclusion Criteria:

* Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study (according to the Thalidomide product/prescribing information).
* Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study (according to the Thalidomide product information).
* Any condition that confounds the ability to interpret data from the study (includes conditions that may affect the absorption of thalidomide, such as gastric bypass surgery, colon resection, etc.).
* Pregnant or lactating females.
* Any surgical or medical conditions that might significantly alter the absorption of study drug, such as gastrectomy, gastroenterostomy, bowel resection, pancreatic injury, or pancreatitis. (Cholecystecomy and appendectomy are permissible.)
* Use of antimyeloma agents (other than thalidomide) or investigational agents within 7 days before the start of the PK phase.
* Prior history of allergic reactions to thalidomide, thalidomide excipients (as referenced in the IB), or to related drugs (ie, lenalidomide).
* Prior history of malignancies, other than multiple myeloma, unless the subject has been free of the disease for >= 3 years (from the time of signing the ICD). Exceptions include the following:

  1. Basal cell carcinoma of the skin
  2. Squamous cell carcinoma of the skin
  3. Carcinoma in situ of the cervix
  4. Carcinoma in situ of the breast
  5. Incidental histological finding of prostate cancer (TNM stage of T1a or T1b)
* Known human immunodeficiency virus (HIV) or infectious hepatitis (type A, B, or C) positivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-11-07 (Actual); Primary Completion 2015-09-23 (Actual); Study Completion 2015-09-23 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters for plasma thalidomide: Tmax Cmax AUC t1/2 CL/F V/F | predose, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours postdose
  PK blood sampling for a single day (on Day 5)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knight, MD, Study Director — Celgene Corporation
Locations (7):
- France (5):
  - Hopital Augustin Morvan, Brest
  - CHU Grenoble, Grenoble
  - CHRU-Hopital Claude Huriez, Lille
  - CHRU Hopital Bretonneau, Tours
  - CHRU Hopital Brabois, Vandœuvre-lès-Nancy
- United Kingdom (2):
  - Christie Hospital NHS Foundation Trust, Manchester
  - Royal Marsden Hospital, Sutton

REFERENCES:
- [Background] Lund J, Gruber A, Lauri B, Duru AD, Blimark C, Swedin A, Hansson M, Forsberg K, Ahlberg L, Carlsson C, Waage A, Gimsing P, Vangsted AJ, Frolund U, Holmberg E, Gahrton G, Alici E, Hardling M, Mellqvist UH, Nahi H. Lenalidomide versus lenalidomide + dexamethasone prolonged treatment after second-line lenalidomide + dexamethasone induction in multiple myeloma. Cancer Med. 2018 Jun;7(6):2256-2268. doi: 10.1002/cam4.1422. Epub 2018 Apr 19. PMID 29673108